CLINICAL TRIAL: NCT02757560
Title: Mechanisms of Dietary Lipid Induced Insulin Resistance
Brief Title: Dietary Lipid Induced Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 029
Record Dates: First submitted 2015-08-04; First posted 2016-05-02 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Insulin Resistance
Keywords: saturated fat; acute insulin resistance; insulin suppression test; dietary fatty acids
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SFA versus control diet (Experimental): Participants will be randomized in a cross-over design to either a weight-maintaining, nutritionally-balanced American Heart Association based eucaloric control diet or a high calorie 24-hour saturated fatty acids enriched diet. For the control diet participants will follow a dietary plan for 72 hours prior to testing. For the SFA diet, participants will be provided with high caloric liquid shakes for breakfast, lunch, dinner and a bedtime snack. On the morning of each test day, participants will be admitted in the fasting state and will provided with a breakfast meal corresponding to the assigned diet (SFA or control). Three hours after completion of the meal, insulin sensitivity will be measured by insulin-suppression test (IST).
  Interventions: Other: SFA diet
- MUFA versus control diet (Experimental): Participants will be randomized in a cross-over design to either a weight-maintaining, nutritionally-balanced American Heart Association based eucaloric control diet or a high calorie 24-hour monounsaturated fatty acids (MUFA) enriched diet. For the control diet participants will follow a dietary plan for 72 hours prior to testing. For the MUFA diet, participants will be provided with high caloric liquid shakes for breakfast, lunch, dinner and a bedtime snack. On the morning of each test day, participants will be admitted in the fasting state and will provided with a breakfast meal corresponding to the assigned diet (MUFA or control). Three hours after completion of the meal, insulin sensitivity will be measured by insulin-suppression test (IST).
  Interventions: Other: MUFA diet
- CARB versus control diet (Experimental): Participants will be randomized in a cross-over design to either a weight-maintaining, nutritionally-balanced American Heart Association based eucaloric control diet or a high calorie 24-hour carbohydrate (CARB) enriched diet. For the control diet participants will follow a dietary plan for 72 hours prior to testing. For the CARB diet, participants will be provided with high caloric liquid shakes for breakfast, lunch, dinner and a bedtime snack. On the morning of each test day, participants will be admitted in the fasting state and will provided with a breakfast meal corresponding to the assigned diet (CARB or control). Three hours after completion of the meal, insulin sensitivity will be measured by insulin-suppression test (IST).
  Interventions: Other: CARB diet

INTERVENTIONS:
Other: SFA diet — SFA versus control diet
  Arms: SFA versus control diet
Other: MUFA diet — MUFA versus control diet
  Arms: MUFA versus control diet
Other: CARB diet — CARB versus control diet
  Arms: CARB versus control diet

SUMMARY:
The overall goal of the proposal is to use a saturated fatty acid (SFA)- enriched, high fat diet to rapidly induce insulin resistance (IR) to provide insight into underlying proximal mechanisms of reduced insulin signaling. Specifically, investigators will identify the initial changes in metabolite concentrations/or pathway signaling ("pathways" will be used to broadly refer to these mechanism specific measures) and therefore the mechanisms most likely responsible for the development of IR during this high fat nutritional challenge. Investigators have assembled a multidisciplinary team that is versed with dietary studies, fatty acid metabolism, measurement of IR and potential mechanisms and mediators of IR, and has experience working with monocytes and the two tissues, muscle and adipose tissue, that are particularly relevant for understanding the effects of high fat diets on IR.

DETAILED DESCRIPTION:
In the first aim, investigators will test whether a short-term high SFA-diet induces and increases insulin resistance in participants with normal and abnormal glucose tolerance, respectively, and determine the associated changes in muscle, adipose tissue and inflammatory cell composition, pathway activation and insulin signaling. Investigators will identify changes in specific signal pathways within these tissues and cells that are hypothesized to mediate or modulate insulin action. Primary mechanisms and pathways examined will include local tissue and systemic inflammation, formation of bioactive lipid intermediates, generation of endoplasmic reticulum (ER) stress, and mitochondrial dysfunction/reactive oxygen formation. By performing studies in participants with normal glucose tolerance and in those with abnormal glucose tolerance investigators will also determine whether the extent and mechanisms of insulin resistance vary with initial degrees of glucose intolerance.

In the second aim, to determine if the extent and mechanisms of insulin resistance vary with dietary composition, investigators will determine whether diets of similar caloric content as the SFA-diet, but enriched in monounsaturated fatty acids or carbohydrates, also induce insulin resistance and whether similar or different mechanistic pathways are responsible. Identifying similarities and differences between diets in inflammatory cell and tissue changes and comparing their relationships with peripheral and tissue insulin action will further clarify which cell and tissue events are most closely linked to development of insulin resistance.

In the final aim, to identify the temporal sequence of mechanistic pathways for insulin resistance and the role of cell and tissue cross-talk in these events, investigators will evaluate inflammatory cell, skeletal muscle and adipose tissue composition and pathway changes after acute, subacute, and more chronic dietary challenges in the same individuals. This will also permit assessment of whether repeated dietary challenges create changes in tissues that resemble those found in more chronic and advanced states of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) from 25-35 kg/m2
* normal glucose tolerance (NGT) diagnosis based on fasting glucose value 100mg/dl and 2 hr glucose <140 mg/dl after a standard 75 gm glucose load; impaired fasting glucose (IFG) on fasting glucose value ≥100 and <126 mg/dl and 2 hr glucose <140 mg/dl; impaired glucose tolerance (IGT) based on 2 hr glucose ≥140 and <200 mg/dl and a fasting glucose <126 mg/dl
* Fasting triglyceride levels <500 mg/dl

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus or a hemoglobin A1c value ≥ 6.5 mg/dl
* Any diabetes medications in the past month, thiazolidinedione medications in the prior 3 months or prior regular use of insulin
* Use of diets, medications (e.g., steroids, weight loss medications ) or current or planned behavior changes (e.g. acute weight loss, exercise training) that will influence changes in IR
* Creatinine >2.0 mg/dl or other laboratory evidence of significant active disease, including hepatic enzyme elevation >2x normal and anemia, known "Nonalcoholic Fatty Liver Disease", bleeding risk
* Malabsorption of fat or other nutrients, severe lactose intolerance or other significant gastrointestinal or pancreatic problems, or recent history of nausea or vomiting
* Acute bacterial or viral illness or evidence of other active infection in the past 4 weeks
* Cardiovascular event, stable or unstable angina or other major illness in the past 6 months
* Current regular use of anti-inflammatory medications (e.g. salicylates > 1 gm/ day) or antioxidants in excess of a daily multi-vitamin, including supplements (e.g. fish oils)
* Lipid lowering medications must be at a stable dose for at least 2 months prior to participation
* Ethanol consumption more than 4 oz day; more than occasional smoker
* Reproductively active women not on contraceptives
* Known allergies, prior reactions or contraindications to proposed clinical agents (e.g Octreotide)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Steady-state plasma glucose (SSPG) | 150-180 min
  Average plasma glucose concentrations during min 150-180 of the insulin suppression test (IST)

SECONDARY OUTCOMES:
Acylcarnitine species | Overnight fast, 3-hour post breakfast
  Measured by chromatography electrospray ionization mass spectrometry on plasma and skeletal muscle samples.
Diacylglycerol species | Overnight fast, 3-hour post breakfast
  Measured on plasma, skeletal muscle and subcutaneous adipose tissue samples.
Ceramides species | Overnight fast, 3-hour post breakfast
  Measured on plasma, skeletal muscle and subcutaneous adipose tissue samples.
Insulin signaling proteins | Overnight fast, 3-hour post breakfast
  Measured on skeletal muscle and subcutaneous adipose tissue samples.
Inflammation markers | Overnight fast, 3-hour post breakfast
  Cytokines and adipokines will be measured in plasma after the diet treatments by ELISA techniques. Mononuclear cells inflammatory gene expression will be measured by real time polymerase chain reaction (RT-PCR). Inflammation will be measured in muscle and adipose tissue by RT-PCR and Western blood analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Principal Investigator — Phoenix Veterans Affairs Health Care System
Locations (1):
- Carl T. Hayden VA Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Subject to VA regulation.